CLINICAL TRIAL: NCT03717220
Title: Reconstructive of Multiple-digit Soft-tissue Defects Using Regional Dorsal Digital Flaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSChen13476
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-06

CONDITIONS: Finger Injuries
Keywords: soft-tissue defects; dorsal branch of the digital artery; regional flap
MeSH Terms: conditions — Finger Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- flaps (Other): flap transferring is used for reconstruction of multiple small-to-moderate soft-tissue defects
  Interventions: Procedure: flap transferring

INTERVENTIONS:
Procedure: flap transferring — we use regional dorsal digital flaps for simultaneous reconstruction of multiple-digit soft-tissue defects

SUMMARY:
Reconstruction of soft-tissue defects in multiple digits poses a significant challenge. This article reports simultaneous reconstruction of multiple small-to-moderate soft-tissue defects using regional dorsal digital island flaps and evaluated the efficacy of their application in such complex situation. A retrospective study will be conducted with 26 patients who had multiple-digit soft-tissue defects treated with regional dorsal digital island flaps. At the final follow-up, we will evaluate the efficacy of their application in such complex situation.

DETAILED DESCRIPTION:
For the recipient where sensory restoration is important, sensation of the flaps is assessed using static two-point discrimination (2PD) and Semmes-Weinstein monofilament (SWM) testing at final follow-up. The cold intolerance of the injured finger is measured using the self-administered Cold Intolerance Severity Score questionnaire that was rated into mild, moderate, severe, and extreme (0-25, 26-50, 51-75 and 76-100). The pain of the injured finger is given subjectively by the patient using a grading system that included grade 1, none; grade 2, mild, no interference with daily activities; grade 3, moderate, patient works but has some limitation in use of the hand because of pain; and grade 4, severe, cannot work or use hand. To sum up, patients report their satisfaction with functional recovery of the injured finger according to the Michigan Hand Outcomes Questionnaire that was based on a 5-point response scale.

ELIGIBILITY:
Inclusion Criteria:

* the separate soft tissue defects with exposed bone or tendon in different digits
* the soft-tissue defect≥1.5 cm and ≤3.5 cm in length
* necessity to preserve digit length
* local tissue near the defect can be used as the donor
* a patient between 15 and 60 years of age

Exclusion Criteria:

* concomitant injuries to the dorsum of the injured finger
* a defect < 1.5 cm and>3.5 cm in length
* a finger degloving injury
* the defect of the thumb

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-07-15 (Actual); Primary Completion 2016-05-10 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Static 2PD test | 18 months to 24 months
  We use a Disk-Criminator to test two nearby points when touching the flap

REFERENCES:
- [Background] Chen C, Tang P, Zhang L, Li X, Zheng Y. Repair of multiple finger defects using the dorsal homodigital island flaps. Injury. 2013 Nov;44(11):1582-8. doi: 10.1016/j.injury.2013.05.019. Epub 2013 Jun 28. PMID 23810451